CLINICAL TRIAL: NCT03797937
Title: Microbiome Benchmarking to Identify Perturbations in Multiple Sclerosis II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Marie D'hooghe, Prof. Dr., National MS Center Melsbroek
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018BDM2
Record Dates: First submitted 2018-03-05; First posted 2019-01-09 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multiple sclerosis (MS) patients (Experimental): Patients will undergo magnetic resonance imaging (MRI). Stool and blood samples will be collected.
  Interventions: Other: Magnetic resonance imaging (MRI)
- Healthy controls (No Intervention): Healthy controls will not undergo magnetic resonance imaging (MRI). Stool and blood samples will be collected.
- Multiple sclerosis (MS) patients undergoing a relapse (No Intervention): Multiple sclerosis (MS) patients undergoing a relapse will not undergo magnetic resonance imaging (MRI). Stool and blood samples will be collected.
- Multiple sclerosis (MS) patients from multiplex MS families (No Intervention): Multiple sclerosis (MS) patients from multiplex MS families will not undergo magnetic resonance imaging (MRI). Stool and blood samples will be collected.

INTERVENTIONS:
Other: Magnetic resonance imaging (MRI) — MRI scanner
  Arms: Multiple sclerosis (MS) patients

SUMMARY:
The goal of this longitudinal study is to (1) explore the association between the gut microbiota and inflammatory disease activity in early onset multiple sclerosis, (2) investigate whether/how gut microbial composition vary when patients experience a relapse, and (3) to assess whether the gut microbiota shows increased similarities between affected pairs of first-degree relatives within the same family when compared with discordant pairs of first-degree relatives.

DETAILED DESCRIPTION:
Using metagenomics, as well as clinical, immunological, and radiological observations, the investigators will investigate if active relapsing-remitting multiple sclerosis patients have a more pro-inflammatory gut microbiota signature than multiple sclerosis patients with less active disease and matched healthy controls.

More specifically, the investigators will investigate whether temporal variability of the gut microbiota is related to inflammatory disease activity in multiple sclerosis, whether changes in the gut microbiota are predictive of future inflammatory disease activity in multiple sclerosis, and whether gut microbiota characteristics are predictive of the disease course after 2 years.

ELIGIBILITY:
Inclusion Criteria patients:

* Diagnosis of MS (as defined by the 2010 McDonald criteria).
* Occurrence of symptoms no longer than 5 years before baseline.
* Aged 18-65.
* Willingness to participate in the study and to sign the informed consent.

Exclusion Criteria patients:

* Treatment with high doses of systemic steroids 2 months before baseline.
* Use of antibiotics 3 months before baseline.
* Chronic gastrointestinal disease (e.g. inflammatory bowel disease, colon cancer).
* Other immune-mediated or autoimmune diseases (e.g. rheumatoid arthritis, diabetes type 1 and 2, psoriasis).

Additional inclusion criteria for MS patients undergoing a relapse:

• Ability to provide a faecal sample within 4 weeks from onset of the first symptoms suggestive of a relapse, before cortisone treatment. A relapse is defined by a new clinical sign or clinical worsening of a previous sign/symptom persisting for >=24 hours in the absence of fever.

Additional exclusion criteria for MS patients undergoing a relapse:

* Treatment with cortisone before collection of baseline faecal sample.
* Evidence of a relapse less than 2 months before baseline.
* Switching disease modifying treatment less than 2 months before baseline.

Inclusion criteria healthy controls:

* Willingness to participate to the study and to sign the informed consent.
* Aged >=18.

Exclusion criteria healthy controls:

* Neurodegenerative disorders.
* Chronic gastrointestinal disease (e.g. inflammatory bowel disease, colon cancer) or autoimmune diseases (e.g. rheumatoid arthritis, diabetes type 1, psoriasis).
* Use of antibiotics 3 months before baseline.
* Treatment with high doses of systemic steroids 2 months before baseline.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical evidence for active disease | 3 years
  Time to first relapse (after baseline) will be reported for all patients.

SECONDARY OUTCOMES:
Radiological evidence for active disease | 3 years
  Occurrence of new contrast-enhancing T1 hyper intense lesions, or changes in white matter lesion volume (i.e. new or enlarging T2 hyper intense lesions)

CONTACTS AND LOCATIONS:
Overall Officials: Marie D'hooghe, M.D., Principal Investigator — National MS Center Melsbroek
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - Nationaal Multiple Sclerose Centrum Melsbroek, Melsbroek, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: No